CLINICAL TRIAL: NCT04116541
Title: MegaMOST - A Multicenter, Open-label, Biology Driven, Phase II Study Evaluating the Activity of Anti-cancer Treatments Targeting Tumor Molecular Alterations /Characteristics in Advanced / Metastatic Tumors.
Brief Title: A Study Evaluating the Activity of Anti-cancer Treatments Targeting Tumor Molecular Alterations/Characteristics in Advanced / Metastatic Tumors.
Acronym: MegaMOST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET19-073 (MegaMOST); 2023-510567-35-00 (EU CTIS Number); 2019-001494-88 (EudraCT Number)
Record Dates: First submitted 2019-10-01; First posted 2019-10-04 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Malignant Solid Tumor
Keywords: Metastatic Solid Neoplasm; Advanced Solid Tumor; Genomic alteration; Targeted therapy; Cabozantinib; Ribociclib; HDM201; Alectinib; Trametinib; Dabrafenib; Avapritinib
MeSH Terms: conditions — Neoplasm Metastasis | interventions — siremadlin; Cohort Studies; ribociclib; cabozantinib; alectinib; regorafenib; trametinib; dabrafenib; avapritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- HDM201 + Ribociclib (Experimental): Patient with documented amplification of Cyclin-dependent kinase 6 (CDK6) and/or Cyclin-dependent kinase 4 (CDK4), and/or cyclin dependent kinase inhibitor 2A (CDKN2A) homozygous deletion, and/or amplification of Cyclin D1 (CCND1) and/or Cyclin D3 (CCND3) with no deletion/losses more than single copy of retinoblastoma 1 (RB1) by copy number and P53 wild-type detected on tumor sample from primary tumor or metastatic lesion.
  Interventions: Drug: HDM201; Drug: Ribociclib
- Cabozantinib (Experimental): Patient with AXL, MET, vascular endothelial growth factor receptor (VEGFR), vascular endothelial growth factor (VEGF), RET, ROS1, MER, Tropomyosin receptor kinase B (TRKB),TIE-2 and/or Tyro3 activating mutations and/or amplification, and/or NTRK translocation and/or ROS1 translocation, and/or MET translocation detected on tumor sample from primary tumor or metastatic lesion.
  Interventions: Drug: Cabozantinib
- Alectinib (Experimental): Activating ALK alterations: translocation, or selected mutations,), or activating rearrangements following validation by central molecular tumor board of Centre Léon Bérard.
  Interventions: Drug: Alectinib
- Regorafenib (Experimental): Patient with Activating mutation and/or amplification and/or rearrangement of VEGFR1-3, TIE-2, KIT, RET, RAF1, BRAF (other than V600 mutations), CRAF, HRAS , PDGFR, FGFR1-2, FLT3 and/or CSF1R, and/or amplification of the ligands, and/or biallelic inactivation of SMAD4, following validation by central molecular tumor board of Centre Léon Bérard.
  Interventions: Drug: Regorafenib
- Trametinib (Experimental): Patient with activating mutation and/or amplification of KRAS (except all KRAS G12 mutations), NRAS, HRAS and/or Mitogen-Activated Protein Kinase Kinase (MAP2K); and/or biallelic inactivation of Neurofibromin 1 (NF1); and/or activating mutation Protein Tyrosine Phosphatase Non-Receptor Type 11 (PTPN11); and/or amplification or translocation of BRAF ; and/or translocation RAF1
  Interventions: Drug: Trametinib
- Trametinib + Dabrafenib (Experimental): Patient with BRAF V600 mutation
  Interventions: Drug: Trametinib; Drug: Dabrafenib
- Avapritinib (Experimental): Activating mutations of KIT exon 17 or PDGFRA exon 18 associated or not to mutation on KIT exon 11 or PDGFRA exon 12/14
  Interventions: Drug: Avapritinib

INTERVENTIONS:
Drug: HDM201 — HDM201 120mg, Every 3 weeks, Per os
  Other Names: Closed cohort
  Arms: HDM201 + Ribociclib
Drug: Ribociclib — Ribociclib 200mg/day, once daily 2 weeks on/1 week off, Per os
  Other Names: Closed cohort
  Arms: HDM201 + Ribociclib
Drug: Cabozantinib — Cabozantinib, 60 mg /day, continuous, Per os
  Other Names: Open cohort
  Arms: Cabozantinib
Drug: Alectinib — Alectinib, 600mg twice daily, Per os
  Other Names: Open cohort
  Arms: Alectinib
Drug: Regorafenib — Regorafenib 160mg, once daily, 3 weeks on/1 week off, Per os
  Other Names: Closed cohort
  Arms: Regorafenib
Drug: Trametinib — Trametinib 2 mg/day, continuous, Per os
  Other Names: Closed cohort
  Arms: Trametinib; Trametinib + Dabrafenib
Drug: Dabrafenib — Dabrafenib 150 mg twice daily, Per os
  Other Names: Open cohort
  Arms: Trametinib + Dabrafenib
Drug: Avapritinib — 300 mg/day,continuous, Per os
  Other Names: Open cohort
  Arms: Avapritinib

SUMMARY:
This trial is a multicenter, open-label, biology driven, phase II study using a sequential Bayesian design, aiming to assess the efficacy and safety of different Matched Targeted Therapy (MTT) in independent and parallel cohorts of treatment.

Patients will be assigned to a treatment cohort based on molecular alterations/characteristics detected on tumor sample from primary tumor or metastatic lesion.

In this protocol, several MTTs treatment cohorts are planned. This study is designed with the flexibility to open new MTTs treatment cohorts and to close existing MTTs treatment cohorts that demonstrate no clinical benefit. Each treatment cohort will be driven separately even though procedures, quality control and reporting, will be common. The protocol will be amended in order to include new treatments or combinations that emerge as being of interest for patients with advanced/metastatic cancers.

All eligible patients will receive study drugs as long as patient experiences clinical benefit in the opinion of the investigator, or until unacceptable toxicity, or until symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status, or withdrawal of consent.

Patients will be permitted to continue study treatment after progressive disease according to RECIST v1.1 if they meet all of the following criteria and following validation of the Sponsor:

* Evidence of clinical benefit as assessed by the investigators,
* Absence of symptoms and signs (including worsening of laboratory values; e.g., new or worsening hypercalcemia) that indicate unequivocal progression of disease,
* No decline in ECOG Performance Status (PS) that can be attributed to disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged of at least 18 years on day of signing informed consent.
* Patients with histologically confirmed diagnosis of metastatic disease or unresectable locally advanced malignancy that is resistant or refractory to standard therapies or for which standard therapies does not exist or is/are not considered appropriate by the investigator.
* A multidisciplinary molecular board must have recommended the specific MTT based on the following documented actionable alterations:

  * Cohort HDM201-Ribociclib : amplification of CDK6 and/or CDK4, and/or CDKN2A homozygous deletion, and/or amplification of CCND1 and/or CCND3 with no deletion/losses more than single copy of RB1 by copy number and P53 wild-type.
  * Cohort Cabozantinib : AXL, MET, VEGFR, VEGF, RET, ROS1, MER, TRKB, TIE-2 and/or Tyro3 activating mutations and/or amplification, and/or NTRK translocation and/or ROS1 translocation, and/or MET translocation.
  * Cohort Alectinib : Activating ALK alterations: translocation, or selected mutations, or activating rearrangements following validation by central molecular tumor board of Centre Léon Bérard.
  * Cohort Regoranib : Activating mutation and/or amplification and/or rearrangement of VEGFR1-3, TIE-2, KIT, RET, RAF1, BRAF (other than V600 mutations), CRAF, HRAS, PDGFR, FGFR1-2, FLT3 and/or CSFR1, and/or amplification of the ligands, and/or biallelic inactivation of SMAD4, following validation by central molecular tumor board of Centre Léon Bérard.
  * Cohort Trametinib : Activating mutation and/or amplification of KRAS (except all KRAS G12 mutations), NRAS, HRAS and/or MAP2K; and/or biallelic inactivation of NF1; and/or activating mutation PTPN11; and/or amplification or translocation of BRAF, and/or translocation RAF1
  * Cohort Trametinib + Dabrafenib : BRAF V600 mutation.
  * Cohort Avapritinib : Activating mutations of KIT exon 17 or PDGFRA exon 18 associated or not to mutation on KIT exon 11 or PDGFRA exon 12/14
* Previously treated by at least one prior line of treatment in the advanced/metastatic setting except for specific tumor type with no standard treatment approved and reimbursed in France following sponsor approval.
* Documented radiological disease progression as per RECIST v1.1 and presence of at least one measurable lesion according to RECIST 1.1 criteria based on screening tumor assessment.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Adequate organ function
* Adequate cardiovascular function
* Specific toxicities related to any prior anti-cancer therapy must have resolved to grade ≤1 , except for alopecia (all grades), grade 2 neuropathy or anemia.
* Unless infertility is proven, men must agree to use effective contraception
* Women of child-bearing potential must have a negative serum pregnancy test within 7 days of first dose of study drug and agree to use effective contraception
* Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study procedures as per protocol.
* Patient must be covered by a medical insurance.

Exclusion Criteria:

* Patients amenable to therapy with curative intent.
* Patients participating to another clinical trial with a medicinal product.
* Patients previously treated with similar MTT meaning any agent targeting the same signaling pathways components.
* Patients unable to swallow oral medication.
* Patients with known hypersensitivity to excipients
* Patients with symptomatic central nervous system (CNS) metastasis who are neurologically unstable or require increasing doses of corticosteroids or local CNS-directed therapy to control their CNS disease.
* Patients with secondary malignancy unless this malignancy is not expected to interfere with the evaluation of study endpoints and is approved by the sponsor. Examples of the latter include: basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, localized prostate cancer, prior malignancy and no evidence of recurrence for ≥ 2 years.
* Patients using, or requirement to use while on the study, or not respecting the minimal wash-out period of medications
* Any clinically significant and/or uncontrolled medical disease that could compromise the patient's ability to tolerate study drug or would likely interfere with study procedures or results.
* Patients with known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Patients who are pregnant or breastfeeding women or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through after the last dose of trial treatment (depanding on cohort).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Estimated)
Dates: Start 2020-01-28 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Progression free rate after 3 months (12 weeks) of treatment | 3 months (12 weeks)
  The proportion of patients with a complete response (CR), a partial response (PR) or a stable disease (SD) at 3 months (12 weeks).

SECONDARY OUTCOMES:
Objective response rate after 3 months (12 weeks) of treatment | 3 months (12 weeks)
  The proportion of patients with a complete or a partial response (CR or PR) as best overall response at 3 months (12 weeks).
Duration of Response | Up to 3 years
  Duration of response applies only to patients whose best overall response was a complete response or a partial response (CR or PR). It will be defined as the time from the date of first documented response (CR or PR) to the date of the first documented progression or death due to underlying cancer and censored at the date of the last adequate tumor assessment.
Progression Free Survival | Up to 3 years
  The time from the date of the first study drug administration to the first documented progression according to investigator assessment of RECIST version 1.1 or death due to any cause
Overall survival | Up to 3 years
  The time from the date of the first study drug administration to the date of death due to any cause
Percentage of long-term responders (> 6 months) | 6 months
  The proportion of long term responders (> 6 months)
Adverse Events | Up to 3 years
  Nature, frequency and severity of Adverse Events (AEs), Serious Adverse Events (SAEs) and Suspected Unexpected Serious Adverse Reactions (SUSARs) graded using Common Terminology Criteria for Adverse Events (CTCAE) V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves BLAY, MD, Principal Investigator — Centre Leon Berard
Locations (10):
- France (10):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine LACASSAGNE, Nice
  - Institut Curie, Paris
  - Institut de Cancérologie de Strasbourg, Strasbourg
  - CHU Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif